CLINICAL TRIAL: NCT05395650
Title: Cyanocobalamin as Photosensitizing Agent Using to Make Cross-linking to Cornea Collagen in Treatment of Progressive Keratoconus
Brief Title: Cyanocobalamin as Photosensitizing Agent
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: EL Romany Ophthalmics Factory (Industry)
Responsible Party: Principal Investigator, Mina ibrahim shalalpy, R&D Manger, EL Romany Ophthalmics Factory
Other Study IDs: CYHEMG
Record Dates: First submitted 2022-05-25; First posted 2022-05-27 (Actual); Last update posted 2023-02-15 (Actual); Status verified 2023-02

CONDITIONS: Keratoconus
MeSH Terms: conditions — Keratoconus

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
is cyanocobalamin active as Photosensitizing Agent instead of riboflavin ? using cyanocobalamin with mix of external collagen to make crosslinking with cornea collagen to make rigid of cornea

ELIGIBILITY:
Inclusion Criteria:

* - Is 20 years or older Has been diagnosed with Keratoconus; Has no other active ocular disease; Is not pregnant or nursing;

Exclusion Criteria:

* Is under the age of 20 Has best corrected visual acuity outside 20/400; Pregnant or nursing at the time of enrollment in the study;

Ages: 20 Years to 40 Years | Sex: All
Age Groups: Adult
Study Population: primary care
Sampling Method: Non-Probability Sample
Enrollment: 1 (Estimated)
Dates: Start 2023-09-01 (Estimated); Primary Completion 2023-10-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
PRESERVATION of presence of red flare by using slit lamb | Base line
  Cyanocobalamin react with cornea collagen and format red flare

IPD SHARING:
Plan to Share IPD: Undecided